CLINICAL TRIAL: NCT03896152
Title: A Multi-center, Randomized, Open-label, Efficacy, Safety, Pharmacokinetics and Pharmacodynamics Study, Assessing Multiple LNP023 Doses in Adult Patients With Paroxysmal Nocturnal Hemoglobinuria and Active Hemolysis
Brief Title: Efficacy, Safety, Pharmacokinetics and Pharmacodynamics Study, Assessing Multiple LNP023 Doses in Adult Patients With Paroxysmal Nocturnal Hemoglobinuria
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLNP023X2204
Record Dates: First submitted 2019-03-28; First posted 2019-03-29 (Actual); Results first posted 2023-12-18 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Paroxysmal Nocturnal Hemoglobinuria
Keywords: Complement; alternative pathway; paroxysmal nocturnal hemoglobinuria; hemolysis; LNP023; PNH; LDH; hemoglobin; Iptacopan
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal; Hemolysis | interventions — iptacopan

STUDY DESIGN:
Intervention Model Description: Randomized, open label study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LNP023 25 mg bid/100 mg bid (Experimental): Four weeks of treatment with iptacopan 25 mg bid in Period 1 followed by treatment with 100 mg bid in Period 2 and Period 3.
  Interventions: Drug: LNP023
- LNP023 50 mg bid/200 mg bid (Experimental): Four weeks of treatment with iptacopan 50 mg bid in Period 1 followed by treatment with 200 mg bid in Period 2 and Period 3.
  Interventions: Drug: LNP023

INTERVENTIONS:
Drug: LNP023 — approximately 2 year of Treatment with LNP023
  Other Names: iptacopan

SUMMARY:
This was a Phase II randomized, open-label, multicenter, efficacy, safety, pharmacokinetic and pharmacodynamic study assessing four iptacopan doses in adult Paroxysmal nocturnal hemoglobinuria (PNH) patients with active hemolysis who were not on eculizumab or any other complement inhibitor less than 3 months prior to first iptacopan dose. Active hemolysis was defined by a lactate dehydrogenase (LDH) value ≥ 1.5 × ULN.

DETAILED DESCRIPTION:
LNP023 is a novel oral small molecular weight compound, that inhibits alternative complement pathway (AP). Blockade of the AP with oral LNP023 has the potential to prevent both intra - and extravascular hemolysis.

The total study duration from Screening until end of study (EOS) was approximately 28 months. This three-period study included:

* Screening phase: of up to 8 weeks
* Period 1: a 4-week treatment period of iptacopan at the first dose in the assigned sequence
* Period 2: an 8-week treatment period at the second dose in the assigned sequence
* Period 3: an approximate 2-year treatment extension period for patients who responded to iptacopan treatment
* Taper down period of 2 weeks was applicable only for patients discontinuing iptacopan treatment (Week 13 for non-responders or Week 109 for responders who did not enter the rollover extension program (REP) (Study CLNP023C12001B / NCT04747613)). During this taper down period, patients were to receive 25 mg qd (once a day) of iptacopan for 7 days, followed by 10 mg qd for 7 additional days.
* An EOS visit that took place 1 week after the last iptacopan administration for patients not joining the REP. For patients joining the REP, the last treatment visit was the EOS visit.
* A safety follow-up call 30 days after the last administration of iptacopan was performed for patients not joining the REP.

Patients were randomized to Sequence 1 or Sequence 2 in a 1:1 ratio. Sequence 1: Four weeks of treatment with iptacopan 25 mg bid (Twice daily) in Period 1 followed by treatment with 100 mg bid in Period 2 and Period 3. If during Period 1, LDH was not reduced by ≥ 40% from the mean of pretreatment values by Week 2 (Day 15 study visit), the iptacopan dose was to be up-titrated to 100 mg bid (starting from Study Day 17). If LDH was not reduced by ≥ 40% from the mean of pretreatment values at Week 4 (Day 29), the iptacopan dose was to be up-titrated to 200 mg bid in Period 2 and Period 3 (starting from Study Day 30). In the approximate 2-year treatment extension (Period 3), patients maintained the same treatment regimen as used in Period 2.

Sequence 2: Four weeks of treatment with iptacopan 50 mg bid in Period 1 followed by treatment with 200 mg bid in Period 2 and Period 3. If during Period 1, LDH was not reduced by ≥ 40% from the mean of pretreatment values by Week 2 (Day 15 study visit), the iptacopan dose was to be up-titrated to 200 mg bid (starting from Study Day 17). In the approximate 2-year treatment extension (Extension Period 3), patients remained on 200 mg bid. No further up-titration was possible

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent must be obtained before any assessment is performed.
2. Male and female patients at least 18 years old at baseline.
3. Diagnosis of active PNH based on documented clone size of ≥10% by RBCs and/or granulocytes, measured by GPI-deficiency on flow cytometry (screening or medical history data acceptable).
4. LDH values > 1.5 x upper limit of the normal range (ULN) for at least 3 measurements over a maximum of 8 weeks prior to Day 1 (Screening, baseline or medical history data acceptable).
5. Hemoglobin level < 10.5 g/dL at Baseline.
6. For Period 3 of the study, patients who as per judgment of Investigator benefit from LNP023 treatment based on reduced hemolytic parameters as compared to Screening and Baseline.
7. Vaccinations against N. meningitidis, S. pneumoniae and H. influenzae is required at least 4 weeks prior to first dosing with LNP023 (existing vaccinations should provide effective titers at time of LNP023 treatment start). If LNP023 treatment has to start earlier than 4 weeks post vaccination, prophylactic antibiotic treatment must be initiated.
8. Able to communicate well with the investigator, to understand and comply with the requirements of the study. -

Exclusion Criteria:

1. Participation in any other investigational drug trial or use of other investigational drugs at the time of enrollment, or within 5 elimination half-lives of enrollment, or within 30 days, whichever is longer; or longer if required by local regulations.
2. Patients treated with eculizumab or any other complement inhibitor less than 3 months prior to study Day 1
3. Known or suspected hereditary or acquired complement deficiency.
4. History of currently active primary or secondary immunodeficiency.
5. History of splenectomy.
6. History of bone marrow/ hematopoietic stem cell or solid organ transplants (e.g. heart, lung, kidney, liver).
7. Evidence of malignant disease, or malignancies diagnosed within the previous 5 years.
8. Patients with laboratory evidence of bone marrow failure (reticulocytes < 60x10E9/L, or platelets < 50x10E9/L or neutrophils < 1x10E9/L) verified both at screening and baseline.
9. History of recurrent meningitis, history of meningococcal infections despite vaccination, as verified at both screening and baseline.
10. Presence or suspicion (based on judgment of the investigator) of active infection within 2 weeks prior to first dose of LNP023, or history of severe recurrent bacterial infections.
11. A positive HIV, Hepatitis B (HBV) or Hepatitis C (HCV) test result at screening.
12. Patients on immunosuppressive agents such, as but not limited to, cyclosporine, tacrolimus, mycophenolate or mycophenolic acid, cyclophosphamide, methotrexate or IV immunoglobulins, less than 8 weeks prior to first treatment with LNP023, unless on a stable regimen for at least 3 months prior to first LNP023 dose.
13. Systemic corticosteroids unless on a stable dose for at least 4 weeks before randomization.
14. Severe concurrent co-morbidities not amenable to active treatment; e.g., patients with severe kidney disease (CKD stage 4, dialysis), advanced cardiac disease (NYHA class IV), severe pulmonary arterial hypertension (WHO class IV), or unstable thrombotic event, as judged by the investigator, both at screening and baseline (unless baseline was skipped).
15. Any medical condition deemed likely to interfere with the patient's participation in the study, or likely to cause serious adverse events during the study.
16. History of hypersensitivity to the study treatment or its excipients or to drugs of similar chemical classes.
17. Female patients who are pregnant or breastfeeding, or intending to conceive during the course of the study.
18. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception during dosing and for 1 week after stopping of investigational drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2019-04-05 (Actual); Primary Completion 2020-04-07 (Actual); Study Completion 2022-02-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- Novartis Investigative Site, Kota Kinabalu, Sabah, Malaysia
- Novartis Investigative Site, Singapore, Singapore
- Novartis Investigative Site, Seoul, South Korea
- Novartis Investigative Site, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com.

REFERENCES:
- [Result] Jang JH, Wong L, Ko BS, Yoon SS, Li K, Baltcheva I, Nidamarthy PK, Chawla R, Junge G, Yap ES. Iptacopan monotherapy in patients with paroxysmal nocturnal hemoglobinuria: a 2-cohort open-label proof-of-concept study. Blood Adv. 2022 Aug 9;6(15):4450-4460. doi: 10.1182/bloodadvances.2022006960. PMID 35561315
- See also: Patient Lay Trial Summary — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=1457

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in 5 investigative sites in 4 countries
Pre-assignment Details: Participants underwent a screening period of up to 8 weeks
Period: Overall Study
Arm/Group | LNP023 25 mg Bid/100 mg Bid | LNP023 50 mg Bid/200 mg Bid
Started | 7 | 6
Completed | 4 | 4
Not Completed | 3 | 2
Not completed — Patient/guardian decision | 1 | 1
Not completed — Adverse Event | 0 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Technical problems | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LNP023 25 mg Bid/100 mg Bid | LNP023 50 mg Bid/200 mg Bid | Total
Number analyzed (Participants) | 7 | 6 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.4 (15.27) | 42.5 (11.98) | 38.2 (13.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 5 | 7
  Male | 5 | 1 | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 7 | 6 | 13

OUTCOME MEASURES:

1. Primary Outcome: Summary of Lactate Dehydrogenase (LDH) Responders
Description: A responder was defined as a patient with at least 60% reduction in LDH compared to Baseline or LDH below the upper limit of normal at any time up to and including Week 12 for that patient.
Time Frame: Week 2, week 4, week 8 and week 12
Population: The overall number of participants analyzed represents the participants in the PD analysis set who had at least one valid measurement of LDH.
  The Pharmacodynamic (PD) analysis set is defined as patients with available PD data, who received any study drug and with no protocol deviations with relevant impact on PD data.
  The number analyzed per row represents the participants with a valid LDH value for that particular visit.
Measure: Count of Participants; unit: Participants
Arm/Group | LNP023 25 mg Bid/100 mg Bid | LNP023 50 mg Bid/200 mg Bid
Number analyzed (Participants) | 7 | 5
Participants
  Responders at week 2 | 6 | 5
  Responders at week 4 | 7 | 5
  Responders at week 8 | 7 | 5
  Responders at week 12 | 7 | 5

2. Secondary Outcome: Percent Change From Baseline in LDH Levels
Description: LDH was used as a hemolysis marker to determine the dose-response effect of iptacopan on the reduction of Paroxysmal nocturnal hemoglobinuria (PNH)-associated hemolysis.
  Active hemolysis is defined by an LDH value ≥ 1.5x upper limit of normal (ULN) Baseline LDH was calculated as the average of the last three screening values prior to randomization.
  Serum was used to calculate the LDH values
Time Frame: Baseline, week 2, week 4, week 8 and week 12
Population: The overall number of participants analyzed represents the participants in the PD analysis set who had at least one valid measurement of LDH.
  The number analyzed per row represents the participants with a valid LDH value at both baseline and that particular visit.
Measure: Mean (Standard Deviation); unit: Percent change in LDH levels
Arm/Group | LNP023 25 mg Bid/100 mg Bid | LNP023 50 mg Bid/200 mg Bid
Number analyzed (Participants) | 7 | 5
Percent change in LDH levels
  Week 2 | -76.52 (18.478) | -84.98 (8.186)
  Week 4 | -79.75 (16.025) | -89.72 (5.430)
  Week 8 | -81.73 (22.832) | -88.30 (8.744)
  Week 12: number analyzed (Participants) | 6 | 4
  Week 12 | -86.17 (8.896) | -85.92 (9.013)

3. Secondary Outcome: Change From Baseline in Hemoglobin
Description: Hemoglobin was used as a hemolysis marker to determine the dose-response effect of iptacopan on the reduction of PNH-associated hemolysis. Whole blood was used to calculate the hemoglobin values.
Time Frame: Baseline, Week 2, week 4, week 8 and week 12
Population: The overall number of participants analyzed represents the participants in the PD analysis set who had at least one valid measurement of hemoglobin.
  The number analyzed per row represents the participants with a valid hemoglobin value both baseline and that particular visit.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | LNP023 25 mg Bid/100 mg Bid | LNP023 50 mg Bid/200 mg Bid
Number analyzed (Participants) | 7 | 4
g/L
  Week 2 | 6.88 (5.812) | 31.83 (10.362)
  Week 4: number analyzed (Participants) | 6 | 4
  Week 4 | 9.61 (11.857) | 36.58 (17.875)
  Week 8 | 15.02 (9.154) | 38.08 (25.956)
  Week 12: number analyzed (Participants) | 6 | 3
  Week 12 | 23.36 (14.378) | 37.11 (26.171)

4. Secondary Outcome: Change From Baseline in Free Hemoglobin
Description: Free hemoglobin was used as a hemolysis marker to determine the dose-response effect of iptacopan on the reduction of PNH-associated hemolysis.
  Whole blood was used to calculate the hemoglobin values.
Time Frame: Baseline, Week 2, week 4, week 8 and week 12
Population: The overall number of participants analyzed represents the participants in the PD analysis set who had at least one valid measurement of free hemoglobin.
  The number analyzed per row represents the participants with a valid free hemoglobin value both at baseline and that particular visit.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | LNP023 25 mg Bid/100 mg Bid | LNP023 50 mg Bid/200 mg Bid
Number analyzed (Participants) | 6 | 4
mg/dL
  Week 2: number analyzed (Participants) | 5 | 3
  Week 2 | -39.84 (26.521) | -13.53 (5.093)
  Week 4 | -31.88 (35.314) | -29.26 (24.218)
  Week 8 | -31.85 (27.517) | -16.31 (48.877)
  Week 12: number analyzed (Participants) | 5 | 2
  Week 12 | -39.58 (31.612) | -14.75 (6.293)

5. Secondary Outcome: Change From Baseline in Carboxyhemoglobin
Description: Carboxyhemoglobin was used as a marker of intravascular and extravascular hemolysis to assess the effect of iptacopan.
  Whole blood was used to calculate the carboxyhemoglobin values.
Time Frame: Baseline, Week 2, week 4, week 8 and week 12
Population: The overall number of participants analyzed represents the participants in the PD analysis set who had at least one valid measurement of carboxyhemoglobin.
  The number analyzed per row represents the participants with a valid carboxyhemoglobin value both at baseline and that particular visit
Measure: Mean (Standard Deviation); unit: Percentage of carboxyhemoglobin
Arm/Group | LNP023 25 mg Bid/100 mg Bid | LNP023 50 mg Bid/200 mg Bid
Number analyzed (Participants) | 7 | 5
Percentage of carboxyhemoglobin
  Week 2 | -0.01 (0.516) | -0.72 (0.697)
  Week 4 | -0.36 (0.472) | -0.98 (0.582)
  Week 8 | -0.50 (0.664) | -1.12 (0.916)
  Week 12: number analyzed (Participants) | 6 | 5
  Week 12 | -0.95 (0.316) | -0.78 (1.704)

6. Secondary Outcome: Change From Baseline in Absolute Reticulocyte Count (ARC)
Description: Reticulocyte count was used as a marker of intravascular and extravascular hemolysis to assess the effect of iptacopan.
  Whole blood was used to calculate the absolute reticulocyte count.
Time Frame: Baseline, week 2, week 4, week 8 and week 12
Population: The overall number of participants analyzed represents the participants in the PD analysis set who had at least one valid measurement of reticulocyte count.
  The number analyzed per row represents the participants with a valid reticulocyte count value both at baseline and that particular visit
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | LNP023 25 mg Bid/100 mg Bid | LNP023 50 mg Bid/200 mg Bid
Number analyzed (Participants) | 7 | 5
10^9 cells/L
  Week 2 | -83.00 (78.750) | -94.23 (112.649)
  Week 4: number analyzed (Participants) | 6 | 5
  Week 4 | -118.44 (76.736) | -132.63 (91.109)
  Week 8 | -113.71 (72.300) | -119.43 (117.048)
  Week 12: number analyzed (Participants) | 6 | 4
  Week 12 | -93.00 (93.425) | -84.92 (123.408)

7. Secondary Outcome: Red Blood Cell Count: Change From Baseline in Erythrocytes
Description: Erythrocytes were used as a marker of intravascular and extravascular hemolysis to assess the effect of iptacopan.
  Whole blood was used to calculate erythrocytes values.
Time Frame: Baseline, week 2, week 4, week 8 and week 12
Population: The overall number of participants analyzed represents the participants in the PD analysis set who had at least one valid measurement of erythrocytes.
  The number analyzed per row represents the participants with a valid erythrocytes value both at baseline and that particular visit.
Measure: Mean (Standard Deviation); unit: 10^12 cells/L
Arm/Group | LNP023 25 mg Bid/100 mg Bid | LNP023 50 mg Bid/200 mg Bid
Number analyzed (Participants) | 7 | 5
10^12 cells/L
  Week 2 | 0.49 (0.194) | 1.02 (0.407)
  Week 4: number analyzed (Participants) | 6 | 5
  Week 4 | 0.74 (0.401) | 1.26 (0.619)
  Week 8 | 1.16 (0.396) | 1.38 (0.796)
  Week 12: number analyzed (Participants) | 6 | 4
  Week 12 | 1.38 (0.531) | 1.38 (0.770)

8. Secondary Outcome: Change From Baseline in C3 Fragment Deposition on PNH RBC
Description: C3 fragment deposition on paroxysmal nocturnal hemoglobinuria red blood cell (PNH RBC) was used as a marker of intravascular and extravascular hemolysis to assess the effect of iptacopan. Accumulation of C3 fragments on red blood cells make them prone to phagocytosis causing extravascular hemolysis.
  Whole blood was used to calculate C3 fragment deposition on PNH RBC values.
Time Frame: Baseline, week 2, week 4, week 8 and week 12
Population: The overall number of participants analyzed represents the participants in the PD analysis set who had at least one valid measurement of C3 fragment deposition.
  The number analyzed per row represents the participants with a valid C3 fragment deposition value both at baseline and that particular visit.
Measure: Mean (Standard Deviation); unit: % C3 fragment deposition on PNH RBC
Arm/Group | LNP023 25 mg Bid/100 mg Bid | LNP023 50 mg Bid/200 mg Bid
Number analyzed (Participants) | 6 | 5
% C3 fragment deposition on PNH RBC
  Week 2 | -1.31 (0.932) | -1.88 (1.457)
  Week 4 | -1.43 (1.217) | -2.74 (2.584)
  Week 8 | -1.85 (1.293) | -2.90 (2.654)
  Week 12: number analyzed (Participants) | 6 | 4
  Week 12 | -1.65 (1.221) | -2.75 (3.002)

9. Secondary Outcome: Mean Haptoglobin Levels
Description: Haptoglobin levels were used as a hemolysis marker to determine the effect of iptacopan on the reduction of PNH-associated hemolysis.
  Serum was used to calculate haptoglobin levels.
Time Frame: Baseline, week 2, week 4, week 8 and week 12
Population: The overall number of participants analyzed represents the participants in the PD analysis set who had at least one valid measurement of haptoglobin.
  The number analyzed per row represents the participants with a valid haptoglobin value for that particular visit.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | LNP023 25 mg Bid/100 mg Bid | LNP023 50 mg Bid/200 mg Bid
Number analyzed (Participants) | 7 | 6
g/L
  Baseline | 0.05 (0.000) | 0.05 (0.000)
  Week 2: number analyzed (Participants) | 7 | 5
  Week 2 | 0.27 (0.251) | 0.41 (0.499)
  Week 4: number analyzed (Participants) | 7 | 5
  Week 4 | 0.24 (0.255) | 0.49 (0.490)
  Week 8: number analyzed (Participants) | 7 | 5
  Week 8 | 0.38 (0.456) | 0.41 (0.374)
  Week 12: number analyzed (Participants) | 6 | 5
  Week 12 | 0.25 (0.356) | 0.18 (0.225)

10. Secondary Outcome: Change From Baseline in Total Bilirubin
Description: Bilirubin levels were used as a hemolysis marker to determine the effect of iptacopan on the reduction of PNH-associated hemolysis.
  Serum was used to calculate bilirubin levels.
Time Frame: Baseline, week 2, week 4, week 8 and week 12
Population: The overall number of participants analyzed represents the participants in the PD analysis set who had at least one valid measurement of bilirubin.
  The number analyzed per row represents the participants with a valid bilirubin value both at baseline and that particular visit.
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | LNP023 25 mg Bid/100 mg Bid | LNP023 50 mg Bid/200 mg Bid
Number analyzed (Participants) | 7 | 5
umol/L
  Week 2 | -19.81 (7.855) | -23.93 (16.735)
  Week 4 | -19.95 (10.620) | -25.93 (15.992)
  Week 8 | -20.24 (12.612) | -25.53 (16.471)
  Week 12: number analyzed (Participants) | 6 | 4
  Week 12 | -21.61 (5.998) | -23.17 (18.195)

11. Secondary Outcome: Mean Platelets Count
Description: Platelet counts were used as a marker of intravascular and extravascular hemolysis to assess the effect of iptacopan.
  Whole blood was used to calculate platelets count.
Time Frame: Baseline, week 2, week 4, week 8 and week 12
Population: The overall number of participants analyzed represents the participants in the PD analysis set who had at least one valid measurement of platelets count.
  The number analyzed per row represents the participants with a valid platelets count value for that particular visit.
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | LNP023 25 mg Bid/100 mg Bid | LNP023 50 mg Bid/200 mg Bid
Number analyzed (Participants) | 7 | 6
10^9 cells/L
  Baseline | 190.45 (59.938) | 156.42 (52.321)
  Week 2: number analyzed (Participants) | 7 | 5
  Week 2 | 223.71 (76.707) | 158.20 (62.683)
  Week 4: number analyzed (Participants) | 6 | 5
  Week 4 | 203.17 (68.520) | 138.20 (57.085)
  Week 8: number analyzed (Participants) | 7 | 5
  Week 8 | 184.43 (50.856) | 141.20 (46.569)
  Week 12: number analyzed (Participants) | 6 | 4
  Week 12 | 189.33 (54.617) | 140.75 (59.618)

12. Secondary Outcome: Mean Ferritin Levels
Description: Ferritin levels were used as a marker of intravascular and extravascular hemolysis to assess the effect of iptacopan.
  Serum was used to calculate ferritin levels.
Time Frame: Baseline, Week 4, Week 8 and week 12
Population: The overall number of participants analyzed represents the participants in the PD analysis set who had at least one valid measurement of ferritin.
  The number analyzed per row represents the participants with a valid ferritin value for that particular visit.
Measure: Mean (Standard Deviation); unit: ug/L
Arm/Group | LNP023 25 mg Bid/100 mg Bid | LNP023 50 mg Bid/200 mg Bid
Number analyzed (Participants) | 7 | 6
ug/L
  Baseline | 176.97 (404.254) | 258.90 (418.114)
  Week 4: number analyzed (Participants) | 7 | 5
  Week 4 | 174.21 (431.042) | 287.88 (517.901)
  Week 8: number analyzed (Participants) | 7 | 5
  Week 8 | 178.31 (443.346) | 304.74 (521.535)
  Week 12: number analyzed (Participants) | 6 | 5
  Week 12 | 203.22 (454.296) | 320.40 (526.783)

13. Secondary Outcome: Mean Clone Size
Description: PNH clone size was used as a marker of intravascular and extravascular hemolysis to assess the effect of iptacopan.
  Whole blood was used to calculate clone size values.
Time Frame: Baseline, week 2, week 4, week 8 and week 12
Population: The overall number of participants analyzed represents the participants in the PD analysis set who had at least one valid measurement of clone size.
  The number analyzed per row represents the participants with a valid clone size value for that particular visit.
Measure: Mean (Standard Deviation); unit: Percentage of PNH Red Blood Cells
Arm/Group | LNP023 25 mg Bid/100 mg Bid | LNP023 50 mg Bid/200 mg Bid
Number analyzed (Participants) | 7 | 6
Percentage of PNH Red Blood Cells
  Baseline: number analyzed (Participants) | 6 | 6
  Baseline | 33.63 (18.149) | 49.13 (29.701)
  Week 2 | 54.95 (12.943) | 65.65 (29.279)
  Week 4 | 65.88 (12.907) | 73.74 (24.616)
  Week 8 | 79.62 (14.308) | 85.06 (16.381)
  Week 12: number analyzed (Participants) | 6 | 4
  Week 12 | 82.87 (11.903) | 91.08 (7.842)

14. Secondary Outcome: Pharmacokinetics Profile: Maximum Plasma Concentration (Cmax)
Description: Cmax is the maximum (peak) observed plasma drug concentration after single dose administration (mass x volume-1).
  PK parameters were determined, using non-compartmental method(s) with Phoenix WinNonlin (Version 8.3), from the plasma concentration-time data.
Time Frame: Day 29 and 57
Population: The overall number of participants analyzed represents the participants in the PK analysis set who had at least one valid measurement of Cmax.
  The Pharmacokinetic (PK) analysis set is defined as patients with at least one available valid PK concentration measurement, who received any study drug and with no protocol deviations that impact on PK data.
  The number analyzed per row represents the participants with a valid Cmax value for that particular visit.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- LNP023 25 mg Bid: Four weeks of treatment with iptacopan 25 mg bid in Period 1
- LNP023 50 mg Bid: Four weeks of treatment with iptacopan 50 mg bid in Period 1
- LNP023 100 mg Bid: treatment with iptacopan 100 mg bid in Period 2 and Period 3.
- LNP023 200 mg Bid: Treatment with iptacopan 200 mg bid in Period 2 and Period 3.
Arm/Group | LNP023 25 mg Bid | LNP023 50 mg Bid | LNP023 100 mg Bid | LNP023 200 mg Bid
Number analyzed (Participants) | 6 | 5 | 6 | 5
ng/mL
  Day 29: number analyzed (Participants) | 6 | 5 | 0 | 0
  Day 29 | 1240 (372) | 1800 (368) |  |
  Day 57: number analyzed (Participants) | 0 | 0 | 6 | 5
  Day 57 |  |  | 2640 (590) | 4520 (1520)

15. Secondary Outcome: Pharmacokinetics Profile: Area Under the Curve Tau (AUCtau)
Description: The AUCtau is the area under the plasma concentration-time curve calculated to the end of a dosing interval (tau) at steady-state (amount x time x volume-1).
  AUCtau was estimated by imputing the 12-hour iptacopan plasma concentration as the PK profile's corresponding pre-dose (0-hour) value, that is, by assuming that at steady-state the iptacopan plasma concentration is the same as the beginning (pre-dose) and end (12 hours postdose) of the dosing interval.
  PK parameters were determined, using non-compartmental method(s) with Phoenix WinNonlin (Version 8.3), from the plasma concentration-time data.
Time Frame: Days 29 and 57
Population: The overall number of participants analyzed represents the participants in the PK analysis set who had at least one valid measurement of AUCtau.
  The number analyzed per row represents the participants with a valid AUCtau value for that particular visit.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | LNP023 25 mg Bid | LNP023 50 mg Bid | LNP023 100 mg Bid | LNP023 200 mg Bid
Number analyzed (Participants) | 6 | 5 | 6 | 5
h*ng/mL
  Day 29: number analyzed (Participants) | 6 | 5 | 0 | 0
  Day 29 | 9630 (3870) | 15200 (2390) |  |
  Day 57: number analyzed (Participants) | 0 | 0 | 6 | 5
  Day 57 |  |  | 19800 (4900) | 33300 (8830)

16. Secondary Outcome: Pharmacokinetics Profile: Minimum Plasma Concentration (Cmin)
Description: Cmin is the lowest plasma concentration observed during a dosing interval at steady state [mass / volume].
  PK parameters were determined, using non-compartmental method(s) with Phoenix WinNonlin (Version 8.3), from the plasma concentration-time data.
Time Frame: Days 29 and 57
Population: The overall number of participants analyzed represents the participants in the PK analysis set who had at least one valid measurement of Cmin.
  The number analyzed per row represents the participants with a valid Cmin value for that particular visit.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | LNP023 25 mg Bid | LNP023 50 mg Bid | LNP023 100 mg Bid | LNP023 200 mg Bid
Number analyzed (Participants) | 6 | 5 | 6 | 5
ng/mL
  Day 29: number analyzed (Participants) | 6 | 5 | 0 | 0
  Day 29 | 520 (299) | 809 (239) |  |
  Day 57: number analyzed (Participants) | 0 | 0 | 6 | 5
  Day 57 |  |  | 931 (460) | 1510 (416)

17. Secondary Outcome: Pharmacokinetics Profile: Time to Reach Maximum Plasma Concentration (Tmax)
Description: Tmax is the time to reach maximum (peak) plasma drug concentration after single dose administration (time).
  PK parameters were determined, using non-compartmental method(s) with Phoenix WinNonlin (Version 8.3), from the plasma concentration-time data.
Time Frame: Days 29 and 57
Population: The overall number of participants analyzed represents the participants in the PK analysis set who had at least one valid measurement of Tmax.
  The number analyzed per row represents the participants with a valid Tmax value for that particular visit.
Measure: Median (Full Range); unit: hours
Arm/Group | LNP023 25 mg Bid | LNP023 50 mg Bid | LNP023 100 mg Bid | LNP023 200 mg Bid
Number analyzed (Participants) | 6 | 5 | 6 | 5
hours
  Day 29: number analyzed (Participants) | 6 | 5 | 0 | 0
  Day 29 | 1.50 [1.00 to 4.00] | 2.00 [1.00 to 2.00] |  |
  Day 57: number analyzed (Participants) | 0 | 0 | 6 | 5
  Day 57 |  |  | 1.53 [0.830 to 2.00] | 2.00 [1.00 to 4.13]

18. Secondary Outcome: Mean Fibrinogen Levels
Description: Fibrinogen level was used as a marker associated with risk of thrombosis. Plasma was used to calculate fibrinogen levels.
Time Frame: Baseline, week 2, week 4, week 8 and week 12
Population: The overall number of participants analyzed represents the participants in the PD analysis set who had at least one valid measurement of fibrinogen.
  The number analyzed per row represents the participants with a valid fibrinogen value for that particular visit.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | LNP023 25 mg Bid/100 mg Bid | LNP023 50 mg Bid/200 mg Bid
Number analyzed (Participants) | 7 | 6
g/L
  Baseline | 3.44 (0.851) | 3.50 (1.178)
  Week 2: number analyzed (Participants) | 7 | 5
  Week 2 | 3.27 (0.935) | 2.93 (0.445)
  Week 4: number analyzed (Participants) | 7 | 5
  Week 4 | 2.80 (0.338) | 2.78 (0.566)
  Week 8: number analyzed (Participants) | 7 | 5
  Week 8 | 2.77 (0.399) | 3.19 (0.531)
  Week 12: number analyzed (Participants) | 6 | 4
  Week 12 | 2.94 (0.802) | 3.09 (0.699)

19. Secondary Outcome: Mean Prothrombin Time (PT)
Description: Prothrombin time was used as a marker associated with risk of thrombosis. Plasma was used to calculate prothrombin time.
Time Frame: Baseline, week 2, week 4, week 8 and week 12
Population: The overall number of participants analyzed represents the participants in the PD analysis set who had at least one valid measurement of prothrombin time.
  The number analyzed per row represents the participants with a valid prothrombin time value for that particular visit.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | LNP023 25 mg Bid/100 mg Bid | LNP023 50 mg Bid/200 mg Bid
Number analyzed (Participants) | 7 | 6
seconds
  Baseline | 10.04 (0.474) | 9.84 (0.210)
  Week 2: number analyzed (Participants) | 7 | 5
  Week 2 | 10.51 (0.426) | 10.18 (0.179)
  Week 4: number analyzed (Participants) | 7 | 5
  Week 4 | 10.29 (0.593) | 10.22 (0.311)
  Week 8: number analyzed (Participants) | 7 | 5
  Week 8 | 10.66 (0.665) | 10.98 (1.678)
  Week 12: number analyzed (Participants) | 6 | 4
  Week 12 | 10.33 (0.501) | 10.13 (0.359)

20. Secondary Outcome: Mean Activated Partial Thromboplastin Time (aPTT)
Description: Activated partial thromboplastin time was used as a marker associated with risk of thrombosis.
  Plasma was used to calculate activated partial thromboplastin time.
Time Frame: Baseline, week 2, week 4, week 8 and week 12
Population: The overall number of participants analyzed represents the participants in the PD analysis set who had at least one valid measurement of aPTT.
  The number analyzed per row represents the participants with a valid aPTT value for that particular visit.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | LNP023 25 mg Bid/100 mg Bid | LNP023 50 mg Bid/200 mg Bid
Number analyzed (Participants) | 7 | 6
seconds
  Baseline | 23.63 (2.280) | 23.32 (2.470)
  Week 2: number analyzed (Participants) | 7 | 5
  Week 2 | 25.83 (2.039) | 25.66 (1.454)
  Week 4: number analyzed (Participants) | 7 | 5
  Week 4 | 26.10 (2.156) | 26.46 (1.802)
  Week 8 | 27.04 (2.914) | 26.84 (3.389)
  Week 12: number analyzed (Participants) | 6 | 4
  Week 12 | 26.48 (3.396) | 24.95 (1.279)

21. Secondary Outcome: Mean D-dimer Levels
Description: D-dimer levels were used as a marker associated with risk of thrombosis. Plasma was used to calculate D-dimer levels.
Time Frame: Baseline, week 2, week 4, week 8 and week 12
Population: The overall number of participants analyzed represents the participants in the PD analysis set who had at least one valid measurement of D-dimer.
  The number analyzed per row represents the participants with a valid D-dimer value for that particular visit.
Measure: Mean (Standard Deviation); unit: mg fibrinogen-equivalent unit (FEU)/L
Arm/Group | LNP023 25 mg Bid/100 mg Bid | LNP023 50 mg Bid/200 mg Bid
Number analyzed (Participants) | 7 | 6
mg fibrinogen-equivalent unit (FEU)/L
  Baseline | 0.39 (0.236) | 0.84 (0.345)
  Week 2: number analyzed (Participants) | 7 | 5
  Week 2 | 0.32 (0.230) | 0.49 (0.189)
  Week 4: number analyzed (Participants) | 7 | 5
  Week 4 | 0.29 (0.199) | 0.43 (0.172)
  Week 8: number analyzed (Participants) | 7 | 5
  Week 8 | 0.24 (0.225) | 0.36 (0.215)
  Week 12: number analyzed (Participants) | 6 | 4
  Week 12 | 0.25 (0.184) | 0.31 (0.147)

22. Secondary Outcome: Mean Thrombin Clotting Time
Description: thrombin clotting time was used as a marker associated with risk of thrombosis. Plasma was used to calculate thrombin clotting time.
Time Frame: Baseline, Week 4, Week 8 and Week 12
Population: The overall number of participants analyzed represents the participants in the PD analysis set who had at least one valid measurement of thrombin clotting time.
  The number analyzed per row represents the participants with a valid thrombin clotting time value for that particular visit.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | LNP023 25 mg Bid/100 mg Bid | LNP023 50 mg Bid/200 mg Bid
Number analyzed (Participants) | 7 | 6
seconds
  Baseline | 14.77 (1.994) | 14.83 (0.916)
  Week 4: number analyzed (Participants) | 7 | 5
  Week 4 | 14.93 (0.642) | 15.58 (1.293)
  Week 8: number analyzed (Participants) | 7 | 5
  Week 8 | 14.90 (0.624) | 15.48 (0.923)
  Week 12: number analyzed (Participants) | 5 | 4
  Week 12 | 16.08 (1.530) | 15.35 (0.526)

ADVERSE EVENTS:
Time Frame: Adverse events were reported from first dose of study treatment until end of study treatment plus 7 days post treatment, up to a maximum duration of 115 weeks.
Description: AEs are reported by period.
Groups:
- LNP023 25mg Bid - Period 1: Four weeks of treatment with iptacopan 25 mg bid in Period 1
- LNP023 50mg Bid - Period 1: Four weeks of treatment with iptacopan 50 mg bid in Period 1
- LNP023 100mg Bid - Period 2: Eight weeks of treatment with iptacopan 100 mg bid in Period 2
- LNP023 200mg Bid - Period 2: Eight weeks of treatment with iptacopan 200 mg bid in Period 2
- LNP023 100mg Bid - Period 3: Two years of Extension Treatment with iptacopan 100 mg bid in Period 3
- LNP023 200mg Bid - Period 3: Two years of Extension Treatment with iptacopan 200 mg bid in Period 3
Arm/Group | LNP023 25mg Bid - Period 1 | LNP023 50mg Bid - Period 1 | LNP023 100mg Bid - Period 2 | LNP023 200mg Bid - Period 2 | LNP023 100mg Bid - Period 3 | LNP023 200mg Bid - Period 3
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/6 | 0/7 | 0/5 | 0/7 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/6 | 0/7 | 0/5 | 0/7 | 0/5
Other Adverse Events (participants affected / at risk) | 2/7 | 4/6 | 3/7 | 1/5 | 4/7 | 4/5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LNP023 25mg Bid - Period 1 (N=7) | LNP023 50mg Bid - Period 1 (N=6) | LNP023 100mg Bid - Period 2 (N=7) | LNP023 200mg Bid - Period 2 (N=5) | LNP023 100mg Bid - Period 3 (N=7) | LNP023 200mg Bid - Period 3 (N=5)
Breakthrough haemolysis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Eosinophilia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Haemolysis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1
Autoimmune thyroiditis (Endocrine disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 0 | 2 | 1
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Antinuclear antibody increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 0 | 0 | 1 | 1
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Blood luteinising hormone increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Blood uric acid increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Blood urine present (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1
Haematocrit increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Haemoglobin increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Reverse tri-iodothyronine increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Thyroxine free increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Impaired fasting glucose (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 3 | 0 | 0 | 1 | 1
Chromaturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Nocturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 0 | 1 | 0
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2021-08-03): https://cdn.clinicaltrials.gov/large-docs/52/NCT03896152/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-14): https://cdn.clinicaltrials.gov/large-docs/52/NCT03896152/SAP_001.pdf